CLINICAL TRIAL: NCT03045380
Title: Effect of Video Game Based Physical Activity Training on Upper Extremity Functions, Walking, Balance and Cognitive Functions in Persons With Multiple Sclerosis
Brief Title: Effect of Video Game Based Physical Activity Training in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2996-GOA
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Game based rehabilitation (Experimental): Game based rehabilitation will be administered once a week for 8 weeks.
  Interventions: Other: Game based physical activity training
- Conventional rehabilitation (Active Comparator): Conventional physiotherapy program will be administered once a week for 8 weeks.
  Interventions: Other: Conventional physiotherapy
- No intervention (No Intervention): Waitlist

INTERVENTIONS:
Other: Game based physical activity training — Based on the physical levels of the patients, appropriate games will be selected and video game based physical activity training will be started. Video games will be played with Xbox One with motion sensor (Microsoft) and a 50'' Liquid Crystal Display. Depending on the prognosis of the patients, the grades of the games and types of the games will be changed. A game based physical activity training session takes 30 to 45 minutes. The program will be administered once a week for 8 weeks.
  Arms: Game based rehabilitation
Other: Conventional physiotherapy — A conventional physiotherapy program including balance, upper extremity, and core stabilization exercises will be implemented. A conventional physiotherapy session takes 30 to 45 minutes. The program will be administered once a week for 8 weeks.
  Arms: Conventional rehabilitation

SUMMARY:
The study was designed to investigate the effect of video games based physical activity training on upper extremity functions, walking, balance and cognitive functions in persons with multiple sclerosis (MS). For this aim, the participants with MS will be divided into three groups: game based physical activity training, conventional rehabilitation, and no intervention groups. The experimental groups will receive therapy sessions once a week for 8 weeks. The no intervention group will receive no intervention, they will be assessed at baseline and after 8 weeks.

DETAILED DESCRIPTION:
MS is an inflammatory, demyelinating, and neurodegenerative disease of the central nervous system. The most common clinical signs and symptoms are fatigue, spasticity, affecting mobility, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction.

In order to increase and maintain the quality of life of individuals with MS these disease-related progressive symptoms need to be managed. For this reason, patients need long-term rehabilitation. This situation reduces the motivation of the people over time and makes the continuity of treatment difficult. Developments in rehabilitation technology aim to contribute to the treatment process as well as to increase the active participation of individuals with chronic diseases.

Current literature has shown that video-based physical activity training as non-pharmacological therapy may be an effective method for symptoms such as balance, tremor, fatigue, cognitive functions in persons with MS.

The primary purpose of the study was to examine the effects and persistence of 8-week video games-based physical activity training in MS patients on upper extremity functions, walking, balance, cognitive functions, quality of life, depression and fatigue. The second aim of the study was to investigate the effect and persistence of traditional physiotherapy of 8 weeks on MS patients on upper extremity functions, walking, balance, cognitive functions, quality of life, depression and fatigue. The third aim of the study is to compare the effects of 8-week videogame-based physical activity training and traditional physiotherapy in MS patients.

Volunteers from persons with MS who are in routine control of the MS Outpatient Clinic of Neurology Department, Faculty of Medicine, Dokuz Eylül University will participate in the study. In accordance with the inclusion criteria, 51 patients were randomly assigned to three groups: 17 patients in the game based rehabilitation group, 17 patients in the conventional rehabilitation group and 17 patients in the no intervention group. Based on the physical levels of the patients, appropriate games will be selected and video game based physical activity training will be started. Video games will be played with Xbox One with motion sensor (Microsoft) and a 52'' Liquid Crystal Display. Depending on the prognosis of the patients, the grades of the games and types of the games will be changed. The program will be administered once a week for 8 weeks. A conventional physiotherapy program including balance, upper extremity, and core stabilization exercises will be implemented. Sessions will take 5-10 minutes warm up, 15-20 minutes exercise and 5-10 minute cool down periods. The program will be administered once a week for 8 weeks. No intervention group formed from waitlist will receive no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting or secondary progressive multiple sclerosis
* Able to walk at least 100 meters without resting
* Able to stand for at least half an hour
* Willingness to participate in the study

Exclusion Criteria:

* Neurological disease other than multiple sclerosis
* A relapse during the study
* Having undergone orthopedic surgery involving the foot-ankle, knee, hip, spine, affecting balance
* Serious cognitive or psychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Change from Baseline at 8 weeks
  The Nine-Hole Peg Test measures finger dexterity.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | Baseline
  Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis.
12-Item Multiple Sclerosis Walking Scale | Change from Baseline at 8 weeks
  The 12-item multiple sclerosis walking scale is a self-report measure of the impact of multiple sclerosis on the individual's walking ability.
Timed 25-Foot Walk | Change from Baseline at 8 weeks
  A clinical tool to evaluate patients for quantitative mobility and leg function performance test in a timed, 25 foot walk.
Six-Spot Step Test | Change from Baseline at 8 weeks
  Six-Spot Step Test reflects a complex array of sensori-motor functions, part of which are lower limb strength, spasticity and coordination, as well as balance.
Five Times Sit to Stand Test | Change from Baseline at 8 weeks
  A measure of functional lower limb muscle strength.
Sit-Up Test | Change from Baseline at 8 weeks
  The Sit-Up Test measures strength and endurance of the abdominals and hip-flexor muscles.
Activities-specific Balance Confidence Scale | Change from Baseline at 8 weeks
  Subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness.
Manual Ability Measure-36 | Change from Baseline at 8 weeks
  The Manual Ability Measurement is a questionnaire on perceived ease or difficulty that a persons may experience when performing unilateral and bilateral activities of daily living tasks.
Beck Depression Inventory | Change from Baseline at 8 weeks
  The Beck Depression Inventory is one of the most widely used psychometric tests for measuring the severity of depression.
Modified Fatigue Impact Scale | Change from Baseline at 8 weeks
  The Modified Fatigue Impact Scale assesses the perceived impact of fatigue.
Multiple Sclerosis International Quality of Life Questionnaire | Change from Baseline at 8 weeks
  The Multiple Sclerosis International Quality of Life Questionnaire is a multi-dimensional, self-administered, disease specific quality of life scale.
Brief International Cognitive Assessment for Multiple Sclerosis | Change from Baseline at 8 weeks
  The Brief International Cognitive Assessment for Multiple Sclerosis is an international initiative to recommend and support a cognitive assessment that is brief, practical and universal. It includes tests of mental processing speed and memory.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Therapy and Rehabilitation, Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No